CLINICAL TRIAL: NCT06902662
Title: Clinical Evaluation of Sanghuangporus Sanghuang in Anti-fatigue
Brief Title: Sanghuangporus Sanghuang Supplementation to Improve Anti-Fatigue Performance in Healthy Adults
Acronym: SSMN4-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Chi-Chang Huang, Professor, National Taiwan Sport University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTSUIRB-113-053; NTSU No. 1141031 (Other Grant/Funding Number: National Taiwan Sport University)
Record Dates: First submitted 2025-03-22; First posted 2025-03-30 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Nutritional Supplementation; Physical Performance
Keywords: muscle strength; anaerobic power; Sanghuangporus sanghuang; DEXA; testosterone

STUDY DESIGN:
Intervention Model Description: A 2-arm randomized, double-blind, parallel-group controlled trial comparing SS-MN4 supplementation versus placebo over 42 days.
Who Masked: Participant, Investigator
Masking Description: The study is a double-blind randomized controlled trial. Both participants and investigators are blinded to group assignments. The SS-MN4 and placebo capsules are identical in appearance, taste, and packaging. Randomization and labeling were managed by an independent third party not involved in the study execution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SS-MN4 Group (Experimental): Participants will take 2 capsules of Sanghuangporus sanghuang mycelia (SS-MN4) daily (1000 mg/day) for 42 days.
  Interventions: Dietary Supplement: SS-MN4
- Placebo Group (Placebo Comparator): Participants will take 2 capsules daily of a placebo identical in appearance and taste to the SS-MN4 supplement for 42 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: SS-MN4 — Participants in the SS-MN4 group will take 2 capsules daily containing a total of 1000 mg/day of Sanghuangporus sanghuang mycelia extract for 42 consecutive days. The capsules are identical in appearance to the placebo.
  Arms: SS-MN4 Group
Dietary Supplement: Placebo — Participants in the placebo group will take 2 capsules daily of an inert substance designed to match the SS-MN4 capsules in color, taste, and appearance. The placebo contains no active ingredients and will be taken for 42 consecutive days.
  Arms: Placebo Group

SUMMARY:
This clinical study aims to evaluate the anti-fatigue and muscle performance-enhancing effects of Sanghuangporus sanghuang mycelia (SS-MN4) capsules in healthy adults. As muscle mass and function naturally decline with age or sedentary lifestyle, there is growing interest in nutritional interventions that may help preserve physical performance and reduce fatigue. Sanghuangporus sanghuang, a traditional medicinal fungus, contains bioactive compounds such as hispidin, known for their antioxidant and anti-inflammatory properties.

The study is a randomized, double-blind, placebo-controlled trial involving 60 healthy male participants aged 20 to 35 years with no regular exercise habits. Participants will be randomly assigned to receive either SS-MN4 capsules (1000 mg/day) or a placebo for 42 days. The intervention aims to determine whether SS-MN4 improves exercise performance, muscle strength, and biochemical markers related to fatigue and muscle damage.

Throughout the study, blood samples, urine samples, exercise tests (e.g., anaerobic power, isometric strength), and body composition analyses (DEXA) will be conducted at multiple time points, including before, during, and after the intervention. In addition, intestinal microbiota analysis and nutritional intake records will be included to assess secondary outcomes.

This research will provide scientific evidence for the health benefits of SS-MN4 in reducing exercise-induced fatigue and improving muscle function. The data collected may support future applications for anti-fatigue health food certification in Taiwan and the development of novel functional supplements for global markets.

DETAILED DESCRIPTION:
This study is designed to investigate the efficacy of Sanghuangporus sanghuang mycelia (SS-MN4) capsules in improving anti-fatigue capacity and muscle performance in healthy adult males without regular exercise habits. The clinical trial is based on preclinical studies showing that hispidin-rich SS-MN4 extracts exert protective effects on muscle cells exposed to dexamethasone-induced damage, suggesting potential benefits for preventing muscle fatigue and atrophy.

With muscle mass and strength declining steadily after age 30, sedentary lifestyles can further accelerate sarcopenia, metabolic dysfunction, and poor physical performance. The development of effective functional ingredients to combat fatigue and muscle deterioration is crucial in modern health promotion, especially in aging populations. Sanghuangporus sanghuang is a traditional medicinal fungus with demonstrated antioxidant, anti-inflammatory, and anti-fatigue properties, making it a promising candidate for functional supplementation.

This is a randomized, double-blind, two-arm, placebo-controlled trial. A total of 60 healthy male participants aged 20 to 35 years will be recruited. They will be randomly assigned to one of two groups: the intervention group will receive two SS-MN4 capsules daily (1000 mg/day), and the placebo group will receive identical capsules with inert content. The intervention period will last 42 days, followed by a 4-week follow-up.

Primary outcome measures include changes in biochemical fatigue markers such as creatine kinase (CK), high-sensitivity C-reactive protein (hs-CRP), cortisol, and testosterone. Muscle function and physical performance will be evaluated through anaerobic power testing, isometric mid-thigh pull (IMTP), vertical jump testing, and endurance tests. Blood and urine samples will be collected at multiple time points (pre-intervention, mid-intervention, post-intervention, and during recovery after exhaustive exercise). Muscle damage indicators (e.g., MDA, myoglobin, 3-methylhistidine/creatinine ratio) will also be assessed.

Secondary outcomes include body composition (measured via DEXA), nutritional intake analysis (via the Cofit app and professional nutritionist review), and gut microbiota profiling using 16S rRNA sequencing. All assessments will be conducted in compliance with Taiwan's Ministry of Health and Welfare anti-fatigue health food evaluation guidelines, and supervised by qualified professionals.

The results will provide clinical evidence supporting SS-MN4 as a novel functional ingredient for enhancing exercise performance and reducing fatigue. Findings will be used for potential health food certification applications and for supporting international marketing of SS-MN4 as a scientifically validated supplement.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants aged between 20 and 35 years
* Non-smokers and non-drinkers
* Not currently taking any dietary supplements or medications
* Normal liver and kidney function
* No chronic diseases such as cardiovascular disease
* Willing and able to provide written informed consent
* Able to comply with study procedures and schedule

Exclusion Criteria:

* Current or past diagnosis of any cardiovascular, liver, kidney, or metabolic disease
* Regular use of dietary supplements, sports nutrition products, or energy drinks
* Known food allergies or intolerances, particularly to mushrooms or herbal products
* Engaging in regular resistance or endurance training in the last 6 months
* Currently taking medications that may interfere with study outcomes
* Smoking or alcohol consumption
* Participation in other clinical trials within the last 3 months

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-10-21 (Estimated)

PRIMARY OUTCOMES:
Change in Serum Creatine Kinase (CK) Level | Baseline (Day 0), Day 21, Day 42, and 3/24/48 hours after exhaustive exercise
  Serum CK will be measured to assess muscle damage related to exercise fatigue using automatic biochemical analyzers (Hitachi 7060).
Change in Isometric Mid-Thigh Pull (IMTP) Strength | Baseline (Day 0) and Day 42
  Isometric muscle strength will be evaluated using IMTP racks and force plates (Kistler) to measure maximal force and rate of force development.

SECONDARY OUTCOMES:
Change in Serum Cortisol and Testosterone Levels | Baseline (Day 0), Day 21, Day 42, and 3/24/48 hours post-exercise
  Serum cortisol and testosterone will be measured by ELISA to evaluate physiological stress and hormone response to supplementation and exercise.
Change in Fat-Free Mass Measured by DEXA | Baseline (Day 0) and Day 42
  Body composition will be assessed using dual-energy X-ray absorptiometry (DEXA; Lunar iDXA) to evaluate changes in muscle mass.
Change in Anaerobic Power (Wingate Test) | Baseline (Day 0) and Day 42
  Anaerobic performance will be measured using a cycle ergometer protocol, assessing peak power, mean power, and fatigue index.
Change in 3-Methylhistidine/Creatinine Ratio in Urine | 24 hours post-exhaustive exercise
  The ratio of 3-Methylhistidine to creatinine in urine will be analyzed to evaluate muscle protein breakdown.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Sport University, Graduate Institute of Sports Science, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves a small sample size and is limited to a specific academic-industry collaboration. Data sharing is not included in the original informed consent and ethical approval.

REFERENCES:
- [Background] Lee MC, Hsu YJ, Ho CS, Chang CH, Liu CW, Huang CC, Chiang WD. Evaluation of the Efficacy of Supplementation with Planox(R) Lemon Verbena Extract in Improving Oxidative Stress and Muscle Damage: A Randomized Double-Blind Controlled Trial. Int J Med Sci. 2021 May 3;18(12):2641-2652. doi: 10.7150/ijms.60726. eCollection 2021. PMID 34104096
- [Background] Huang WC, Lee MC, Lee CC, Ng KS, Hsu YJ, Tsai TY, Young SL, Lin JS, Huang CC. Effect of Lactobacillus plantarum TWK10 on Exercise Physiological Adaptation, Performance, and Body Composition in Healthy Humans. Nutrients. 2019 Nov 19;11(11):2836. doi: 10.3390/nu11112836. PMID 31752370